CLINICAL TRIAL: NCT07383571
Title: Safety and Efficacy of Oral Hyoscine Butylbromide Versus Topical EMLA Spray in Reducing Pain During Hysterosalpingography: A Randomized Double-Blind Placebo-Controlled Trial
Brief Title: Oral Hyoscine vs. Topical EMLA vs. Placebo for Pain Reduction During Hysterosalpingography
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Aljazeera Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSG-Analgesia-2025
Record Dates: First submitted 2025-09-21; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Hysterosalpingography
MeSH Terms: interventions — Butylscopolammonium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral Hyoscine butylbromide and Placebo Spray (Experimental)
  Interventions: Drug: Oral Hyoscine butylbromide and Placebo Spray
- Topical EMLA Spray and Placebo Oral Tablet (Active Comparator)
  Interventions: Drug: Topical EMLA Spray and Placebo Oral Tablet
- Double Placebo (Placebo Comparator)
  Interventions: Other: Double Placebo

INTERVENTIONS:
Drug: Oral Hyoscine butylbromide and Placebo Spray — Hyoscine butylbromide 20 mg oral tablet, single dose 30 min before HSG PLUS placebo cervical spray
  Arms: Oral Hyoscine butylbromide and Placebo Spray
Drug: Topical EMLA Spray and Placebo Oral Tablet — EMLA spray (lidocaine 2.5% + prilocaine 2.5%), 3 sprays to ectocervix/external os, 10 min before HSG plus placebo oral tablet
  Arms: Topical EMLA Spray and Placebo Oral Tablet
Other: Double Placebo — oral placebo tablet plus placebo cervical spray
  Arms: Double Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled, will evaluate whether oral hyoscine butylbromide or topical eutectic lidocaine-prilocaine (EMLA) spray reduces pain during hysterosalpingography (HSG) compared with placebo

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled, three-arm clinical trial will evaluate whether oral hyoscine butylbromide or topical eutectic lidocaine-prilocaine (EMLA) spray reduces pain during hysterosalpingography (HSG) compared with placebo

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing HSG for infertility evaluation

Regular cycles; procedure scheduled in proliferative phase (days 6-12)

Negative urine pregnancy test on procedure day

Exclusion Criteria:

* Known hypersensitivity to hyoscine, lidocaine, prilocaine.

Use of systemic analgesics, sedatives, or antispasmodics within 24 hrs pre-HSG

Chronic pelvic pain or severe dysmenorrhea requiring regular analgesics

Active pelvic infection, uterine anomaly, cervical stenosis requiring anesthesia

History of contrast allergy

Inability to cooperate with VAS reporting

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity (VAS) during cervical instrumentation (after tenaculum and cannula placement) | IMMEDIATE(1 MINUTE)
  Pain will be measured using a 0-10 Numerical Rating Scale (NRS), where 0 indicates no pain and 10 indicates the worst pain imaginable
Pain at end of uterine filling | INTRA-PROCEDURE
  "Pain will be measured using a 0-10 Numerical Rating Scale (NRS), where 0 indicates no pain and 10 indicates the worst pain imaginable

SECONDARY OUTCOMES:
Baseline pain after speculum insertion | INTRAPROCEDURE
  "Pain will be measured using a 0-10 Numerical Rating Scale (NRS), where 0 indicates no pain and 10 indicates the worst pain imaginable
pain 30 minutes post procedure | 30 minutes post-procedure
  "Pain will be measured using a 0-10 Numerical Rating Scale (NRS), where 0 indicates no pain and 10 indicates the worst pain imaginable
women satisfaction | 30 minutes postprocedure
  it will be measured using a 0-10 Numerical Rating Scale (NRS) like scale , where 0 indicates no satisfaction and 10 indicates the maximum satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, MD, Principal Investigator — Algazeera Hospital
Locations (1):
- Al Gezeera Hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No